CLINICAL TRIAL: NCT03677492
Title: Cytochalasin D Supplementation to ICSI Handling Medium
Brief Title: Supplementing Intracytoplasmic Sperm Injection Handling Medium With Cytochalasin D ( ICSI-CD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IbnSinaIVF-ICSI-CD
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Cytochalasin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handling Medium Supplemented with Cytochalasin D (Experimental)
  Interventions: Other: Medium Supplemented with Cytochalasin D
- Handling Medium as it is. (No Intervention)

INTERVENTIONS:
Other: Medium Supplemented with Cytochalasin D — A medium with in-house supplementation of Cytochalasin D to decrease oocyte degeneration after ICSI and improve the survival rate
  Arms: Handling Medium Supplemented with Cytochalasin D

SUMMARY:
Vienna Consensus has identified 10% damage rate after ICSI as a competency value. Despite the highest quality embryologists doing ICSI, degeneration sometimes occurs due to oocyte factors such as the fragile membrane, etc. Cytochalasin D serves to facilitate spindle or pronuclear transfer procedures helping to reduce the damage rate with no harm reported. Using Cytochalasin D during ICSI could serve to rescue some oocytes from the degeneration allowing for more chances of viable zygotes.

ELIGIBILITY:
Inclusion Criteria:

* ICSI indicated participants

Exclusion Criteria:

-

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Oocyte survival rate | 6 days of culture

SECONDARY OUTCOMES:
Fertilization rate | 6 days of culture
Blastocyst formation rate | 6 days of culture
Embryo utilization rate | 6 days of culture
Clinical pregnancy rate | three months
Implantation rate | 7 weeks
Ongoing pregnancy rate | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Banon Assiut, Asyut
  - IbnSina IVF Center, IbnSina Hospital, Sohag